CLINICAL TRIAL: NCT06583902
Title: Management of Anaemia in Patients with Infectious Endocarditis Who Are Candidates for Cardiac Surgery: the AMERICA Trial
Brief Title: Management of Anemia in Patients with EndocaRditis Infectious Candidates for Cardiac Surgery: the AMERICA Study
Acronym: AMERICA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 6780
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Erythropoietin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- prospective: Data obtained in patients prospectively included in the study will be compared with those from a retrospective case-control population of patients treated consecutively in the previous two years.
  Interventions: Drug: Intravenous iron
- Retrospective: Data obtained in patients prospectively included in the study will be compared with those from a retrospective case-control population of patients treated consecutively in the previous two years.
  Interventions: Other: Retrospective case-control analysis

INTERVENTIONS:
Drug: Intravenous iron — Patients with an absolute deficiency (ferritin ≤100 μg/L) or functional deficiency (ferritin ≤ 300 μg/L with transferrin saturation ≤20%) receive iron supplementation, through a single administration of an iron preparation for intravenous use administered according to the doses present in the technical data sheet.
  Other Names: erythropoietin
  Groups: prospective
Other: Retrospective case-control analysis — the only routine clinical data collection (Hb, iron status, direct and indirect Coombs test, IL6, erythropoietin dosage, number of units of blood components possibly transfused)
  Groups: Retrospective

SUMMARY:
Infective endocarditis (EI) is an extremely serious disease requiring prolonged hospitalisation, complex management by multidisciplinary teams and high healthcare costs. Anemia is also emerging as a virtually constant condition associated with endocarditis, as evidenced by its inclusion in the variables used to calculate risk scores.Anemia associated with infective endocarditis (EI) has a remarkably complex and multifactorial pathogenesis.It is essential to treat anaemia in patients with EI as an integral part of their overall therapy, in what is now called patient blood management. Blood transfusion is not the only approach available to treat this condition. It is essential to correct any deficiencies, whether iron or vitamins. In addition, some patients may benefit from the administration of erythropoiesis-stimulating agents.

ELIGIBILITY:
Inclusion Criteria: Patients with endocarditis who are candidates for elective surgery; Male and female patients aged > 18 years; Patients who have given written consent to participate in the study and to have their clinical data processed for the purposes of the study.

Exclusion Criteria: Age < 18 years; Patients with hypersensitivity (bronchial asthma, urticaria, allergic phenomena) to preparations of intravenous iron, folic acid, vitamin B12, erythropoietin; Patients who have not given written consent to participate in the study and who have specifically refused the use of their clinical data for the purposes of the study; Patients participating in other investigational trials; Any other clinical condition that in the opinion of the investigator would make the patient unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Foundation for infective endocarditis with an indication for cardiac surgery presenting anaemia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Assessing improvement in anemia and reduction of transfusion support in the study population | 18 months
  To assess the improvement in anaemia and reduction in transfusion support in the study population compared to a selected control population (patients with endocarditis who underwent surgery in the 24 months prior to PBM implementation).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Malattie Infettive, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No